CLINICAL TRIAL: NCT01337804
Title: A Single Dose, Comparative, Open-label, Randomized, Crossover Bioequivalence Study of Omeprazole Administered as Zegerid® Powder for Oral Suspension 20 mg and Prilosec 40 mg Capsule in Healthy Subjects
Brief Title: A Study to Compare Omeprazole Administered as Zegerid® Powder and as Prilosec® Capsule in Healthy Participants (P08050)(CL2010-12)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18136; P08050 (Other: Merck)
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — omeprazole, sodium bicarbonate drug combination; Suspensions; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zegerid-Prilosec (Experimental): Participants receive Zegerid in Period 1 and Prilosec in Period 2, with a 10- to 21-day washout between study drug administrations.
  Interventions: Drug: omeprazole/sodium bicarbonate; Drug: omeprazole magnesium
- Prilosec-Zegerid (Experimental): Participants receive Prilosec in Period 1 and Zegerid in Period 2, with a 10- to 21-day washout between study drug administrations.
  Interventions: Drug: omeprazole/sodium bicarbonate; Drug: omeprazole magnesium

INTERVENTIONS:
Drug: omeprazole/sodium bicarbonate — Single 20 mg dose of omeprazole/sodium bicarbonate powder for oral suspension
  Other Names: Zegerid Powder for Oral Suspension
Drug: omeprazole magnesium — Single 40 mg capsule of omeprazole given orally
  Other Names: Prilosec

SUMMARY:
This study compares the bioequivalence of omeprazole administered as either Zegerid® powder for oral suspension 20 mg or as Prilosec 40 mg capsule to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant is of non-Asian origin.
* Female participants of reproductive potential must have a negative pregnancy test and agree to use (and/or have their partner use) two acceptable methods of birth control beginning at the screening visit, throughout the study, and until 2 weeks after the last dose of study drug.
* Participant has a Body Mass Index (BMI) ≤35 kg/m2 at the screening visit.
* Participant is judged to be in good health.
* Participant has no clinically significant abnormality on electrocardiogram (ECG).
* Participant has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least 6 months.

Exclusion Criteria:

* Participant is mentally or legally incapacitated, has significant emotional problems at the time of screening visit or has a history of a clinically significant psychiatric disorder over the last 5 to 10 years. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Participant has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Participant has taken any gastric antisecretory drugs (e.g., histamine receptor type-2 antagonists [H2RAs] or proton pump inhibitors [PPIs]), antacids, or any other prescription or over- the-counter (OTC) medications within 14 days prior to Period 1 and during the trial.
* Participant has been treated with any trial drug or therapy, or participated in a clinical trial in the 30 days prior to Period 1.
* Participant has any laboratory test result prior to dosing in Period 1 deviating from the normal reference ranges established by the local laboratory by more than 20% that the investigator judges to be of possible clinical significance.
* Participant has an estimated creatinine clearance of ≤80 mL/min based on the Cockcroft-Gault equation.
* Participant has a history of stroke, chronic seizures, or major neurological disorder.
* Participant has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases. Participants with a history of uncomplicated kidney stones or childhood asthma may be enrolled in the study at the discretion of the investigator.
* Participant has a history of neoplastic disease.
* Participant is a nursing mother.
* Participant has any history or serologic evidence of hepatitis B or C with abnormal liver function tests (except for benign, self-limited hepatitis A >5 years prior to randomization), hepatic or biliary tract disease, or a history of gastrointestinal tract surgery.
* Participant has an allergy or hypersensitivity to any component/excipient of the study drugs, has a history of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
* Participant is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort [hypericum perforatum]) beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods), until the telephone follow-up. There may be certain medications that are permitted. Participants must be explicitly warned of the potential risk of taking erythromycin, clarithromycin, nefazodone, ketoconazole, itraconazole, cyclosporine, and human immunodeficiency virus (HIV)protease inhibitors during the study.
* Participant consumes excessive amounts of alcohol, defined as greater than 3 glasses per day of alcoholic beverages (1 glass is approximately equivalent to: 10 ounces of beer, 4 ounces of wine, or 1 ounce of distilled spirits).
* Participant has consumed grapefruit juice, grapefruits and grapefruit products within 2 weeks prior to administration of the initial dose of study drug, and does not agree to refrain from their consumption throughout the study (including the washout interval between treatment periods) and until the telephone follow-up.
* Participant consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, chocolate, or other caffeinated beverages per day.
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 30 days prior to Period 1. The 4-week window will be derived from the date of the last study procedure (i.e., telephone follow-up) in the previous study to the screening visit of the current study.
* Participant is currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year.
* There is any concern by the investigator regarding the safe participation of the participant in the study or for any other reason; the investigator considers the participant inappropriate for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from 0 to infinity (AUC[0-∞]) | Up to 12 hours post-dose
Maximum plasma concentration (Cmax) | Up to 12 hours post-dose